CLINICAL TRIAL: NCT01617564
Title: Paracervical Block (PCB) During II-trimester Abortion- A Randomized Controlled Trial
Brief Title: Paracervical Block During II-trimester Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristina Gemzell Danielsson (Other)
Responsible Party: Sponsor-Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: W2010IM
Record Dates: First submitted 2012-05-31; First posted 2012-06-12 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Second Trimester Medical Abortion
Keywords: medical abortion; second trimester; para cervical blockage; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacain (Active Comparator)
  Interventions: Drug: bipuvacain
- Sodium Chloride (Sham Comparator)
  Interventions: Other: NaCl

INTERVENTIONS:
Drug: bipuvacain — PCB with 20ml bupivakain or sodium cloride 9mg/ml will be administered one hour following misorpostol administration (first dose).
  Other Names: (Marcain® 2,5mg/ml)
  Arms: Bupivacain
Other: NaCl — PCB with 20ml sodium chloride (9mg/ml) inactive (sham) comparator
  Arms: Sodium Chloride

SUMMARY:
Paracervical blockage can reduce severe pain during second trimester induced medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women who request second trimester medical abortion (13-22 weeks gestation according to ultrasound)
* 18 years of age or older
* able to understand and communicate in Swedish
* able to understand the study related information and willing to give her
* informed consent to participation in the study

Exclusion Criteria:

* Known allergy to bupivakain or related substances

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain score | at 24 hours
  Pain indicated on VAS at specific time intervals during the induction to expulsion

SECONDARY OUTCOMES:
Efficacy | after 24h from induction
  Number of complete abortions within 24h without the need for surgery
Time to abortion | at 24hours
  Time from induction (first dose of misoprostol) to expulsion
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at 6 to 8 weeks
  AEs reported during the time period from mifepristone (Day 1)until follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Dept of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm
  - Södersjukhuset, Stockholm

REFERENCES:
- [Derived] Andersson IM, Benson L, Christensson K, Gemzell-Danielsson K. Paracervical block as pain treatment during second-trimester medical termination of pregnancy: an RCT with bupivacaine versus sodium chloride. Hum Reprod. 2016 Jan;31(1):67-74. doi: 10.1093/humrep/dev286. Epub 2015 Nov 15. PMID 26573530